CLINICAL TRIAL: NCT04860622
Title: Normal Range of TSH and FT4 in Pregnancy
Acronym: NRTSHTURKEY
Status: Completed | Type: Observational
Sponsor: Sehit Prof. Dr. Ilhan Varank Sancaktepe Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Arzu Bilge Tekin, Specialist M.D., Sehit Prof. Dr. Ilhan Varank Sancaktepe Training and Research Hospital
Other Study IDs: NR TSH TURKEY
Record Dates: First submitted 2021-04-22; First posted 2021-04-27 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Hypothyroidism; Pregnancy Related; Thyroid; Dysfunction; Iodine Deficiency
Keywords: Hypothyroidism; Pregnancy; trimester; thyroid dysfunction; iodine level
MeSH Terms: conditions — Hypothyroidism; Thyroid Diseases | interventions — Pregnancy Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women: 500 pregnant women with a singleton pregnancy, free of pre-existing thyroid disease, that do not use thyroid interfering medication, that did not undergo IVF treatment, and are TPOAb negative. Serum thyroid function tests will be obtained on the first visit.
  Interventions: Diagnostic Test: Serum thyroid function tests

INTERVENTIONS:
Diagnostic Test: Serum thyroid function tests — At the first hospital visit, the blood tests will be made for TSH, FT4, FT3, and beta HCG concentration measurement
  Other Names: Beta HCG and thyroid peroxidase antibody; Thyroid ultrasonography

SUMMARY:
Physiological changes necessitate the use of pregnancy-specific reference ranges for thyrotrophin (TSH) and free T4 (FT4) to diagnose thyroid dysfunction during pregnancy. Although many centers use fixed upper limits for TSH of 2.5 or 3.0 mU/L, this may lead to overdiagnosis or even overtreatment.

The new guidelines of the American Thyroid Association have considerably changed recommendations regarding thyroid function reference ranges in pregnancy accordingly. Any hospital or physician that is still using the 2.5 or 3.0 mU/l cut-off for TSH during pregnancy should evaluate their own lab-specific cut-offs.

The investigator's objective is to establish a rational reference range of serum TSH for the diagnosis of subclinical hypothyroidism in the first, second, and third trimester of pregnant women in the Sancaktepe region in Turkey.

DETAILED DESCRIPTION:
Serum thyroid function tests (including T3, T4, TSH, Anti-TPO) will be obtained from the singleton pregnancies in the first, second, and third trimester to determine the local specific normal ranges.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Free of pre-existing thyroid disease
* That do not use thyroid interfering medication
* That did not undergo IVF treatment
* TPOAb negative

Exclusion Criteria:

* Adolescent pregnancy
* Patient with pre-existing thyroid disease
* TPOAb positive
* Patient using thyroid interfering medication
* That had IVF treatment

Ages: 18 Years to 50 Years | Sex: Female
Age Groups: Adult
Study Population: Turkish pregnant women living in Sancaktepe Region of Turkey
Sampling Method: Probability Sample
Enrollment: 528 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
TSH | On day 1
  Trimester specific TSH level

SECONDARY OUTCOMES:
free T4 | On day 1
  Trimester specific free T4 level

CONTACTS AND LOCATIONS:
Overall Officials: Murat Yassa, MD, Principal Investigator — Specialist
Locations (1):
- Sehit Prof Dr Ilhan Varank Sancaktepe Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Alexander EK, Pearce EN, Brent GA, Brown RS, Chen H, Dosiou C, Grobman WA, Laurberg P, Lazarus JH, Mandel SJ, Peeters RP, Sullivan S. 2017 Guidelines of the American Thyroid Association for the Diagnosis and Management of Thyroid Disease During Pregnancy and the Postpartum. Thyroid. 2017 Mar;27(3):315-389. doi: 10.1089/thy.2016.0457. PMID 28056690
- [Background] Panesar NS, Li CY, Rogers MS. Reference intervals for thyroid hormones in pregnant Chinese women. Ann Clin Biochem. 2001 Jul;38(Pt 4):329-32. doi: 10.1258/0004563011900830. PMID 11471873
- [Background] Donovan LE, Metcalfe A, Chin A, Yamamoto JM, Virtanen H, Johnson JA, Krause R. A Practical Approach for the Verification and Determination of Site- and Trimester-Specific Reference Intervals for Thyroid Function Tests in Pregnancy. Thyroid. 2019 Mar;29(3):412-420. doi: 10.1089/thy.2018.0439. Epub 2019 Feb 4. PMID 30595114